CLINICAL TRIAL: NCT01080300
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety and Efficacy of Gabapentin Extended Release (G-ER_ Tablets in the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: Breeze3:Study of Gabapentin Extended Release in the Treatment of Vasomotor Symptoms(Hot Flashes)in Postmenopausal Women
Acronym: Breeze3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 81-0064
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Hot Flashes
Keywords: Hot Flushes; Vasomotor Symptoms; Menopausal Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin Extended Release (Experimental): Active treatment
  Interventions: Drug: Gabapentin Extended Release
- Placebo (Other): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin Extended Release — Gabapentin ER 1800mg daily
  Arms: Gabapentin Extended Release
Drug: Placebo — Sugar pill
  Arms: Placebo

SUMMARY:
Depomed's Gabapentin Extended Release is an investigational, extended release formulation of Gabapentin that is being studied for the treatment of Hot Flashes/Hot Flushes in postmenopausal women

DETAILED DESCRIPTION:
The primary study objective is to assess the efficacy of G-ER dosed at 1800mg daily (600mg AM, 1200mg PM), compared to placebo in reducing the average daily frequency and severity score of moderate to severe hot flashes in postmenopausal women at weeks 4 & 12 of the efficacy treatment period, compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women who seek treatment for hot flashes
* Patients using hormone replacement therapy(HRT) must be willing to discontinue treatment
* Patients must be experiencing moderate to severe hot flashes
* Patients must be able to sign the informed consent
* Patients must be able to enter simple commands and complete questionnaires on the frequency and severity of their hot flashes using an electronic diary

Other inclusions apply.

Exclusion Criteria:

* Patients with hypersensitivity to Gabapentin
* Patients with severe chronic diarrhea, chronic constipation, uncontrolled irritable bowel syndrome (IBS) or unexplained weight loss
* Patients treated with estrogen pellets or injectable progestin drug therapy within 6 months.
* Patients currently treated with Gabapentin or Pregabalin for any indication, including vasomotor symptoms

Other exclusions apply.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Sathyanarayana, Study Director — Depomed
Locations (66):
- United States (66):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Berkeley, California
  - Roseville, California
  - San Diego, California
  - Denver, Colorado
  - Danbury, Connecticut
  - Milford, Connecticut
  - Brooksville, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Gainesville, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Decatur, Georgia
  - Idaho Falls, Idaho
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Overland Park, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Paw Paw, Michigan
  - Brooklyn Center, Minnesota
  - Las Vegas, Nevada
  - Reno, Nevada
  - Moorestown, New Jersey
  - Plainsboro, New Jersey
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Wexford, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Goose Creek, South Carolina
  - Greer, South Carolina
  - Rapid City, South Dakota
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Seattle, Washington

REFERENCES:
- [Derived] Pinkerton JV, Kagan R, Portman D, Sathyanarayana R, Sweeney M; Breeze 3 Investigators. Phase 3 randomized controlled study of gastroretentive gabapentin for the treatment of moderate-to-severe hot flashes in menopause. Menopause. 2014 Jun;21(6):567-73. doi: 10.1097/GME.0b013e3182a7c073. PMID 24149930

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 600 subjects were randomly assigned to treatment: 302 in G-ER 1800 mg group and 298 in placebo group. Of these 600 subjects, 595 subjects (300 in G-ER 1800 mg group and 295 in placebo group) received study treatment and were included in the safety population, and 593 subjects were included in the intent-to-treat (ITT) population.
Groups:
- G-ER 1800 mg: Gabapentin extended-release (G-ER) 1800 mg
- Sugar Pill: Placebo 1800 mg
Period: Overall Study
Arm/Group | G-ER 1800 mg | Sugar Pill
Started | 300 (302 subjects were randomized, but only 300 received study treatment.) | 295 (298 subjects were randomized, but only 295 received study treatment.)
Completed | 206 | 191
Not Completed | 94 | 104
Not completed — Adverse Event | 49 | 35
Not completed — Lack of Efficacy | 12 | 15
Not completed — Protocol Violation | 7 | 13
Not completed — Lost to Follow-up | 10 | 6
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 12 | 28
Not completed — Reasons not specified | 4 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | G-ER 1800 mg | Sugar Pill | Total
Number analyzed (Participants) | 299 | 294 | 593
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (6.1) | 54.0 (6.0) | 54.0 (6.1)
Age, Customized [Number; unit: participants]
  < 65 years | 280 | 282 | 562
  >=65 years | 19 | 12 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 294 | 593
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 215 | 197 | 412
  Black | 74 | 82 | 156
  Asian | 1 | 2 | 3
  Hispanic | 9 | 9 | 18
  Other | 0 | 4 | 4
Frequency of hot flashes [Mean (Standard Deviation); unit: hot flashes] — Number of hot flashes in a 24-hour period.
  hot flashes
    Mild | 1.5 (2.8) | 1.5 (3.3) | 1.5 (3.1)
    Moderate | 6.4 (5.3) | 6.1 (4.9) | 6.3 (5.1)
    Severe | 7.1 (10.6) | 6.5 (5.4) | 6.8 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: G-ER at 1800mg Daily Compared With Placebo in Reducing the Average Daily Frequency of Moderate to Severe Hot Flashes at Weeks 4 & 12 of the Efficacy Treatment Period, Compared With Baseline.
Description: G-ER dosed at 1800mg daily(600mg AM, 1200mg PM), compared with placebo in reducing the average daily frequency of moderate to severe hot flashes in post menopausal women at Week 4 of the efficacy treatment period compared with Baseline and at Week 12 of the efficacy treatment period compared with Baseline.
Time Frame: Baseline, Week 4, and Week 12
Population: Intent-to-treat (ITT) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: hot flashes
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
hot flashes
  Baseline LOCF Average Daily Frequency at Week 4 | -6.72 [-7.24 to -6.19] | -5.01 [-5.54 to -4.49]
  Baseline LOCF Average Daily Frequency at Week 12 | -7.64 [-8.21 to -7.07] | -6.50 [-7.07 to -5.94]
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Baseline LOCF Average Daily Frequency at Week 4: Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily number of moderate to severe hot flashes at Week 4; Test type: Superiority or Other; p = 0.0003, Based on Van Eltereen — P-value for the test of difference of the least square mean change from baseline between Gabapentin ER 1800 mg and placebo group is based on the F-test of Type III analysis; Multiplicity addressed by requiring significance for all primary endpoints; Mean Difference (Net) = -1.70, 95% CI 2-sided [-2.31 to -1.09], Standard Error of Mean 0.311 — Based on ANCOVA
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Baseline LOCF Average Daily Frequency at Week 12: Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily number of moderate to severe hot flashes at Week 12; Test type: Superiority or Other; p = 0.1000, Based on Van Elteren — [p-value comment as in outcome 1, analysis 1]; Multiplicity addressed by requiring significance for all primary endpoints; Mean Difference (Net) = -1.14, 95% CI 2-sided [-1.80 to -0.48], Standard Error of Mean 0.335 — Based on ANCOVA

2. Primary Outcome: G-ER at 1800mg Daily Compared With Placebo in Reducing the Average Daily Severity Score of Moderate to Severe Hot Flashes at Weeks 4 & 12 of the Efficacy Treatment Period, Compared With Baseline.
Description: G-ER dosed at 1800mg daily(600mg AM, 1200mg PM), compared with placebo in reducing the average daily severity score of moderate to severe hot flashes in post menopausal women (score defined as "Mild" (1), "Moderate" (2), and "Severe" (3)) at Week 4 of the efficacy treatment period compared with Baseline and at Week 12 of the efficacy treatment period compared with Baseline.
Time Frame: Baseline, Week 4, and Week 12
Population: Intent-to-treat (ITT) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
scores on a scale
  Baseline LOCF Average Daily Severity at Week 4 | -0.42 [-0.51 to -0.33] | -0.22 [-0.31 to -0.13]
  Baseline LOCF Average Daily Severity at Week 12 | -0.65 [-0.77 to -0.52] | -0.46 [-0.58 to -0.34]
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Baseline LOCF Average Daily Severity Score at Week 4: Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily severity score of moderate to severe hot flashes at Week 4; Test type: Superiority or Other; p < 0.0001, Based on Van Elteren — [p-value comment as in outcome 1, analysis 1]; Multiplicity addressed by requiring significance for all primary endpoints; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.31 to -0.10], Standard Error of Mean 0.052 — Based on ANCOVA
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Baseline LOCF Average Daily Severity Score at Week 12: Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily severity score of moderate to severe hot flashes at Week 12; Test type: Superiority or Other; p = 0.0004, Based on Van Elteren — [p-value comment as in outcome 1, analysis 1]; Multiplicity addressed by requiring significance for all primary endpoints; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.33 to -0.04], Standard Error of Mean 0.072 — Based on ANCOVA

3. Secondary Outcome: G-ER at 1800mg Daily Compared With Placebo in Reducing the Average Daily Frequency of Moderate to Severe Hot Flashes at Week 24 of the Efficacy Treatment Period, Compared With Baseline.
Description: G-ER dosed at 1800mg daily(600mg AM, 1200mg PM), compared with placebo in reducing the average daily frequency of moderate to severe hot flashes in post menopausal women at Week 24 of the efficacy treatment period compared with Baseline.
Time Frame: Baseline, Week 24
Population: Completer Population
Measure: Least Squares Mean (95% Confidence Interval); unit: hot flashes
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 185 | 177
hot flashes | -8.99 [-9.71 to -8.27] | -7.91 [-8.62 to -7.19]
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Baseline LOCF Average Daily Frequency at Week 24: Null hypothesis: no treatment differences relative to placebo in mean change from baseline in observed average daily number of moderate to severe hot flashes at Week 24; Test type: Superiority or Other; p = 0.1510, Based on Van Elteren; Multiplicity addressed by requiring significance for all primary endpoints; Mean Difference (Net) = -1.08, 95% CI 2-sided [-1.98 to -0.19], Standard Error of Mean 0.453 — Based on ANCOVA

4. Secondary Outcome: G-ER at 1800mg Daily Compared With Placebo in Reducing the Average Daily Severity Score of Moderate to Severe Hot Flashes at Week 24 of the Efficacy Treatment Period, Compared With Baseline.
Description: G-ER dosed at 1800mg daily(600mg AM, 1200mg PM), compared with placebo in reducing the average daily severity score of moderate to severe hot flashes in post menopausal women (score defined as "Mild" (1), "Moderate" (2), and "Severe" (3)) at Week 24 of the efficacy treatment period compared with Baseline.
Time Frame: Baseline, Week 24
Population: Completer Population
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 185 | 177
scores on a scale | -0.86 [-1.03 to -0.69] | -0.64 [-0.81 to -0.47]
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Baseline LOCF Average Daily Severity Score at Week 24: Null hypothesis: no treatment differences relative to placebo in mean change from baseline in observed average daily severity score of moderate to severe hot flashes at Week 24; Test type: Superiority or Other; p = 0.0004, Van Elteren; Multiplicity addressed by requiring significance for all primary endpoints; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.44 to -0.00], Standard Error of Mean 0.110 — Based on ANCOVA

5. Secondary Outcome: Patient Global Impression of Change (PGIC) Scales at Weeks 12 and 24 of the Efficacy Treatment Period.
Description: Proportion of patients who were categorized as "very much" or "much improved" for PGIC at Week 12 and Week 24. Scale range is 6 categories: "minimum value = very much worse" to "maximum value = very much improved".
Time Frame: Week 12 and Week 24
Population: Intent-to-treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
Participants
  Baseline LOCF Proportion at Week 12 | 173 | 130
  Baseline LOCF Proportion at Week 24 | 156 | 114
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Proportion of patients who were categorized as "very much" or "much improved" in PGIC at Week 12. Null Hypotheses: no treatment differences, relative to placebo in the proportion of patients who were categorized as "very much" or "much improved" in the PGIC score at week 12; Test type: Superiority or Other; p = 0.0008, 2-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 13.6, 95% CI 2-sided [5.7 to 21.6] — Risk difference defined as treatment difference in proportion of responders
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Proportion of patients who were categorized as "very much" or "much improved" in PGIC at Week 24; Test type: Superiority or Other; p = 0.0009, 2-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 13.4, 95% CI 2-sided [5.5 to 21.3] — Risk difference defined as treatment difference in proportion of responders

6. Secondary Outcome: Clinical Global Impression of Change (CGIC) Scales at Weeks 12 and 24 of the Efficacy Treatment Period.
Description: Proportion of patients who were categorized as "very much" or "much improved" in CGIC at Week 12 and Week 24. Scale range is 6 categories: "minimum value = very much worse" to "maximum value = very much improved".
Time Frame: Week 12 and Week 24
Population: Intent-to-treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
Participants
  Baseline LOCF Proportion at Week 12 | 173 | 122
  Baseline LOCF Proportion at Week 24 | 159 | 124
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Proportion of patients who were categorized as "very much" or "much improved" in CGIC at Week 12. Null Hypotheses: no treatment differences, relative to placebo in the proportion of patients who were categorized as "very much" or "much improved" in the CGIC score at week 12; Test type: Superiority or Other; p < 0.0001, 2-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 16.4, 95% CI 2-sided [8.4 to 24.3] — Risk difference defined as treatment difference in proportion of responders
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Week 24; Test type: Superiority or Other; p = 0.0070, 2-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 11.0, 95% CI 2-sided [3.0 to 19.0] — Risk difference defined as treatment difference in proportion of responders

7. Secondary Outcome: Percent of Patients With 75% or Greater Reduction in Average Daily Frequency of Moderate to Severe Hot Flashes
Time Frame: Baseline, Week 12, and Week 24
Population: Intent-to-treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
Participants
  Baseline LOCF Proportion at Week 12 | 125 | 101
  Baseline LOCF Proportion at Week 24 | 146 | 122
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Week 12; Test type: Superiority or Other; p = 0.0609, two-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 7.5, 95% CI 2-sided [-0.3 to 15.2] — Risk difference defined as treatment difference in proportion of responders
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Week 24; Test type: Superiority or Other; p = 0.0720, two-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 7.3, 95% CI 2-sided [-0.7 to 15.3] — Risk difference defined as treatment difference in proportion of responders

8. Secondary Outcome: Percent of Patients With 75% or Greater Reduction in Average Daily Severity Score of Moderate to Severe Hot Flashes
Time Frame: Baseline, Week 12, and Week 24
Population: Intent-to-treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
Participants
  Baseline LOCF Average Daily Score at Week 12 | 48 | 36
  Baseline LOCF Average Daily Score at Week 24 | 62 | 48
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Week 12; Test type: Superiority or Other; p = 0.1825, two-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 3.8, 95% CI 2-sided [-1.8 to 9.4] — Risk difference defined as treatment difference in proportion of responders
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Week 24; Test type: Superiority or Other; p = 0.1662, two-sample Z test; No multiplicity adjustments were made for secondary efficacy outcomes; Risk Difference (RD) = 4.4, 95% CI 2-sided [-1.8 to 10.7] — Risk difference defined as treatment difference in proportion of responders

9. Secondary Outcome: Change From Baseline to Weeks 4, Week 12, and Week 24 in Average Daily Sleep Interference Score.
Description: Sleep Interference Score Range: Minimum value = 0, maximum value = 10 Lower scores indicate better outcome (ie, less interference)
Time Frame: Baseline, Week 4, Week 12, and Week 24
Population: Intent-to-treat (ITT) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
units on a scale
  Change from Baseline to Week 4: LOCF daily rating: number analyzed (Participants) | 297 | 293
  Change from Baseline to Week 4: LOCF daily rating | -2.67 [-3.00 to -2.33] | -1.31 [-1.64 to -0.97]
  Change from Baseline to Week 12: LOCF daily rating: number analyzed (Participants) | 297 | 293
  Change from Baseline to Week 12: LOCF daily rating | -3.09 [-3.47 to -2.71] | -2.17 [-2.56 to -1.79]
  Change from Baseline to Week 24: LOCF daily rating: number analyzed (Participants) | 298 | 293
  Change from Baseline to Week 24: LOCF daily rating | -3.15 [-3.56 to -2.75] | -2.20 [-2.60 to -1.80]
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Change from Baseline to Week 4: LOCF daily sleep interference rating; Test type: Superiority or Other; p < 0.0001, ANCOVA — The P value (versus placebo) for the pairwise test of difference of the LS mean change from Baseline between the G-ER 1800-mg and placebo-treatment groups was based on the F test of type III analysis; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -1.36, 95% CI 2-sided [-1.75 to -0.97], Standard Error of Mean 0.196
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Change from Baseline to Week 12: LOCF daily sleep interference rating; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -0.92, 95% CI 2-sided [-1.36 to -0.47], Standard Error of Mean 0.226
Statistical Analysis 3: Comparison: G-ER 1800 mg vs Sugar Pill; Change from Baseline to Week 24: LOCF daily sleep interference rating; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -0.95, 95% CI 2-sided [-1.42 to -0.49], Standard Error of Mean 0.237

10. Secondary Outcome: Changes From Baseline in Sleep Quality Scores, Measured by the Insomnia Severity Index (ISI) to Week 4, Week 12, and Week 24 of the Efficacy Treatment Period.
Description: Insomnia Severity Index (ISI) scored on 4-point Likert-scales ('0' not at all - '4' extremely) for 7 sub-categories. Final score is sum of each sub-category generating a total sleep quality score (0-28). Minimum value = 0, maximum value = 28 (Lower scores indicate better outcome (ie, less severity)).
Time Frame: Baseline, Week 4, Week 12, and Week 24
Population: Intent-to-treat (ITT) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
scores on a scale
  Change from Baseline to Week 4: LOCF ISI rating: number analyzed (Participants) | 298 | 294
  Change from Baseline to Week 4: LOCF ISI rating | -6.47 [-7.67 to -5.82] | -4.13 [-5.04 to -3.21]
  Change from Baseline to Week 12: LOCF ISI rating: number analyzed (Participants) | 298 | 294
  Change from Baseline to Week 12: LOCF ISI rating | -7.02 [-7.96 to -6.09] | -5.17 [-6.10 to -4.25]
  Change from Baseline to Week 24: LOCF ISI rating: number analyzed (Participants) | 298 | 294
  Change from Baseline to Week 24: LOCF ISI rating | -6.71 [-7.65 to -5.77] | -4.95 [-5.88 to -4.01]
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; Change from Baseline to Week 4: LOCF daily insomnia severity index (ISI) rating; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -2.62, 95% CI 2-sided [-3.67 to -1.56], Standard Error of Mean 0.537
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; Change from Baseline to Week 12: LOCF daily insomnia severity index (ISI) rating; Test type: Superiority or Other; p = 0.0007, ANCOVA — [p-value comment as in outcome 9, analysis 1]; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -1.85, 95% CI 2-sided [-2.92 to -0.78], Standard Error of Mean 0.543
Statistical Analysis 3: Comparison: G-ER 1800 mg vs Sugar Pill; Change from Baseline to Week 24: LOCF daily insomnia severity index (ISI) rating; Test type: Superiority or Other; p = 0.0014, ANCOVA; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -1.76, 95% CI 2-sided [-2.84 to -0.69], Standard Error of Mean 0.548

11. Secondary Outcome: Changes From Baseline in Quality of Life Scores, Measured by the Menopause-Specific Quality of Life Questionnaire (MENQOL) to Weeks, 4, 12, 24 of the Efficacy Treatment Period.
Description: 4 sub-categories each scored individually: Minimum value = 1, maximum value = 8.
  Overall summary score was mean of the 4 sub-category scores (minimum = 1 and maximum = 8).
  Lower scores indicate better outcome (ie, less severity)
Time Frame: Baseline, Week 4, Week 12, and Week 24
Population: Intent-to-treat (ITT) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 299 | 294
scores on a scale
  Baseline LOCF MENQOL score at Week 4: number analyzed (Participants) | 297 | 294
  Baseline LOCF MENQOL score at Week 4 | -0.91 [-1.06 to -0.77] | -0.71 [-0.85 to -0.57]
  Baseline LOCF MENQOL score at Week 12: number analyzed (Participants) | 297 | 294
  Baseline LOCF MENQOL score at Week 12 | -1.01 [-1.16 to -0.87] | -0.87 [-1.01 to -0.72]
  Baseline LOCF MENQOL score at Week 24: number analyzed (Participants) | 297 | 294
  Baseline LOCF MENQOL score at Week 24 | -1.01 [-1.17 to -0.86] | -0.96 [-1.11 to -0.81]
Statistical Analysis 1: Comparison: G-ER 1800 mg vs Sugar Pill; MENQOL score at Week 4; Test type: Superiority or Other; p = 0.0137, ANCOVA — The p-value (vs. Placebo) for the test of difference of the LS mean change from baseline between Gabapentin ER 1800mg and placebo group is based on the F-test of Type III analysis; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.37 to -0.04], Standard Error of Mean 0.084
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; MENQOL score at Week 12; Test type: Superiority or Other; p = 0.0872, ANCOVA — [p-value comment as in outcome 11, analysis 1]; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.31 to 0.02], Standard Error of Mean 0.084
Statistical Analysis 3: Comparison: G-ER 1800 mg vs Sugar Pill; MENQOL score at Week 24; Test type: Superiority or Other; p = 0.5607, ANCOVA — [p-value comment as in outcome 11, analysis 1]; No multiplicity adjustments were made for secondary efficacy outcomes; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.23 to 0.13], Standard Error of Mean 0.091

12. Secondary Outcome: Safety of G-ER Measuring Columbia-Suicide Severity Rating Scale (C-SSRS).
Description: Columbia-Suicide Severity Rating Scale (C-SSRS). Subjects were classified as 0=no suicidal ideation or 1=suicidal ideation. Outcome Measure is number of participants with or without suicidal ideation.
  Higher counts without suicidal ideation = better outcome.
Time Frame: Week 4, Week 12, Week 24/Early Termination, Week 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Extended Release | Placebo
Number analyzed (Participants) | 300 | 295
Participants
  Patients Taking C-SSRS at Week 4: number analyzed (Participants) | 260 | 257
  Patients Taking C-SSRS at Week 4: With Suicidal Ideation | 0 | 0
  Patients Taking C-SSRS at Week 4: Without Suicidal Ideation | 260 | 257
  Patients Taking C-SSRS at Week 12: number analyzed (Participants) | 225 | 215
  Patients Taking C-SSRS at Week 12: With Suicidal Ideation | 1 | 0
  Patients Taking C-SSRS at Week 12: Without Suicidal Ideation | 224 | 215
  Patients Taking C-SSRS at Week 24/EarlyTermination: number analyzed (Participants) | 271 | 267
  Patients Taking C-SSRS at Week 24/EarlyTermination: With Suicidal Ideation | 0 | 1
  Patients Taking C-SSRS at Week 24/EarlyTermination: Without Suicidal Ideation | 271 | 266
  Patients Taking C-SSRS at Week 28: number analyzed (Participants) | 257 | 243
  Patients Taking C-SSRS at Week 28: With Suicidal Ideation | 1 | 0
  Patients Taking C-SSRS at Week 28: Without Suicidal Ideation | 256 | 243

ADVERSE EVENTS:
Time Frame: Adverse events collected for a total of 28-42 weeks: from after signing the informed consent to the end of the study (Week 28).
Description: Adverse event collection began after signing the informed consent and continued through Week 28 visit; serious adverse events followed for 30 days after study completion.
Arm/Group | G-ER 1800 mg | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 4/300 | 7/295
Other Adverse Events (participants affected / at risk) | 102/300 | 53/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER 1800 mg (N=300) | Sugar Pill (N=295)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER 1800 mg (N=300) | Sugar Pill (N=295)
Dizziness (Nervous system disorders) | 38 (44) | 10 (10)
Headache (Nervous system disorders) | 28 (28) | 24 (25)
Somnolence (Nervous system disorders) | 18 (18) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 18 (18) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that sponsor shall have the right to first publication of study results which is intended to be a joint, multi-center publication. Following first publication, the PI may publish study data or results, provided however PI submits proposed publication to sponsor for review at least 60 days prior to the date of proposed publication. Sponsor may remove any information that is considered confidential and/or proprietary other than study data.

ACCEPTED FOR PUBLICATION IN "MENOPAUSE".